CLINICAL TRIAL: NCT07299240
Title: Remote Ischemic Conditioning for Sleep Disturbances and Other Non-motor Symptoms in Parkinson's Disease: a Randomized, Single-blind, Sham-controlled Clinical Study
Brief Title: Remote Ischemic Conditioning for Sleep Disturbances and Other Non-motor Symptoms in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY088-02
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease (PD); Insomnia
Keywords: remote ischemic conditioning; Parkinson's disease; insomnia; non-motor symptoms
MeSH Terms: conditions — Parkinson Disease; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are blinded to group allocation. Active and sham RIC devices are identical in appearance, and both groups undergo the same procedures except for cuff inflation pressure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active RIC group (Experimental): Participants receive active remote ischemic conditioning plus standard antiparkinsonian medications.
  Interventions: Device: Remote ischemic conditioning device
- Sham RIC group (Sham Comparator): Participants receive sham remote ischemic conditioning (low-pressure cuff inflation) plus standard antiparkinsonian medications.
  Interventions: Device: Sham remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning device — An automated upper-limb cuff device is applied to one arm to induce brief episodes of limb ischemia and reperfusion. In the active RIC group, the cuff is inflated to a high pressure (approximately 200 mmHg) sufficient to occlude arterial blood flow, and then deflated repeatedly according to a pre-set program recommended by the manufacturer. RIC is performed twice daily for 7 consecutive days.
  Other Names: RIC training device
  Arms: Active RIC group
Device: Sham remote ischemic conditioning — The same device and procedure are used as in the active RIC group, but the cuff is inflated only to a low pressure (approximately 60 mmHg) that does not occlude arterial blood flow. Sham RIC is performed twice daily for 7 consecutive days.
  Arms: Sham RIC group

SUMMARY:
This single-center, randomized, single-blind, sham-controlled clinical trial aims to evaluate whether remote ischemic conditioning (RIC) can improve sleep disturbances and other non-motor symptoms in patients with Parkinson's disease (PD). Forty-eight PD patients with insomnia will be randomly assigned in a 1:1 ratio to receive either active RIC (cuff inflation to high pressure) or sham RIC (cuff inflation to low pressure) for 7 consecutive days, in addition to their standard antiparkinsonian medications. Subjective sleep scales, sleep diaries, validated rating scales for motor and non-motor symptoms, and overnight polysomnography will be used to assess treatment effects at baseline, after the 7-day intervention, and during short-term follow-up. The study will also explore potential mechanisms of RIC by combining EEG, functional MRI, retinal optical coherence tomography, and blood biomarkers.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disorder characterized not only by motor symptoms, but also by a wide spectrum of non-motor symptoms. Sleep disturbances, including insomnia and fragmented sleep, are highly prevalent in PD and markedly impair quality of life, yet current pharmacological therapies have limited efficacy and may cause adverse effects. Remote ischemic conditioning (RIC) is a non-invasive intervention induced by repeated brief episodes of limb ischemia and reperfusion using an inflatable cuff. Experimental and clinical studies suggest that RIC can modulate immune responses, humoral mediators, neural activity and circadian rhythms. Based on these observations, we hypothesize that RIC may improve sleep disturbances and other non-motor symptoms in PD.

In this study, 48 PD patients with insomnia will be recruited from the outpatient clinics and inpatient wards of Nanjing Brain Hospital. Eligible participants will be randomized (1:1) to an active RIC group or a sham RIC group on top of stable antiparkinsonian medications. Each participant will undergo two nights of polysomnography (one adaptation night and one baseline recording), comprehensive clinical assessments, EEG, retinal optical coherence tomography (OCT) and functional MRI (fMRI) before the intervention. RIC or sham RIC will then be performed twice daily for 7 consecutive days. After completion of the 7-day intervention, polysomnography, EEG, fMRI, OCT, clinical rating scales and blood sampling will be repeated. A further clinical and neurophysiological assessment will be conducted approximately 21 days after the end of RIC to evaluate the persistence of treatment effects. The primary objective is to determine whether RIC improves subjective and objective sleep parameters in PD patients with insomnia. Secondary objectives include assessing changes in other non-motor symptoms, motor symptoms, cognition, mood, autonomic function, quality of life and exploratory imaging and blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease according to the Movement Disorder Society (MDS) clinical diagnostic criteria.
* Age between 50 and 70 years.
* Disease duration ≤ 5 years.
* Hoehn and Yahr stage I-III in the "on" state.
* Presence of insomnia that meets the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria and clinically significant sleep complaints (for example, Parkinson's Disease Sleep Scale-2 [PDSS-2] total score ≥ 18 points).
* On a stable regimen of antiparkinsonian medications for at least 4 weeks prior to enrollment, with no expected dose changes during the study period.
* Able to understand the study procedures and provide written informed consent (or consent provided by a legally authorized representative when appropriate).

Exclusion Criteria:

* Secondary insomnia due to other severe medical conditions (e.g., uncontrolled cardiopulmonary, hepatic, renal, or endocrine diseases).
* Current psychotic symptoms or severe anxiety or depression (e.g., Hamilton Anxiety Scale score ≥ 14 or Hamilton Depression Scale score ≥ 17).
* Other primary sleep disorders such as moderate-to-severe obstructive sleep apnea, restless legs syndrome, periodic limb movement disorder, or rapid eye movement sleep behavior disorder that require specific treatment.
* History of significant cerebrovascular disease, brain tumor, central nervous system infection, or other neurological disorders that may interfere with sleep or study assessments.
* Contraindications to remote ischemic conditioning (RIC), including severe peripheral arterial disease of the upper limbs, local soft tissue infection or damage at the cuff site, subclavian artery thrombosis, malignant hypertension, severe cardiac disease, active bleeding disorders, or other conditions judged unsafe by the investigator.
* Contraindications to MRI or EEG examinations (e.g., pacemaker, severe claustrophobia, metallic implants incompatible with MRI).
* Participation in another interventional clinical trial within the past 3 months.
* Inability to comply with the study procedures or follow-up visits, as judged by the investigator.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Parkinson's Disease Sleep Scale-2 (PDSS-2) total score | From baseline to 7 days after the start of RIC
  The PDSS-2 is a 15-item patient-reported questionnaire assessing sleep problems in Parkinson's disease. Total scores range from 0 to 60, with higher scores indicating more severe sleep disturbances. The primary outcome is the change in PDSS-2 total score from baseline to the end of the 7-day RIC or sham RIC intervention.

SECONDARY OUTCOMES:
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) total score (0-260 points; higher scores indicate worse motor and non-motor symptoms). | Baseline to 7 days after RIC
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is used to assess motor and non-motor symptoms in Parkinson's disease. The total score ranges from 0 to 260 points, with higher scores indicating more severe impairment. The outcome measure is the change in MDS-UPDRS total score from baseline to 7 days after remote ischemic conditioning (RIC).
Change in Montreal Cognitive Assessment (MoCA) total score (0-30 points; higher scores indicate better cognitive function). | Baseline to 7 days after RIC
  The Montreal Cognitive Assessment (MoCA) is a 30-point screening instrument for global cognitive function. Total scores range from 0 to 30 points, with higher scores indicating better cognition. The outcome measure is the change in MoCA total score from baseline to 7 days after remote ischemic conditioning (RIC).

CONTACTS AND LOCATIONS:
Overall Officials: Haochen Sun, Principal Investigator — Department of Neurology, the Affiliated Brain Hospital of Nanjing Medical University
Locations (1):
- the Affiliated Brain Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the main published results will be made available to qualified researchers upon reasonable request and after approval by the principal investigator and the Institutional Review Board.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 5 years after publication of the main results.
Access Criteria: Researchers must submit a methodologically sound proposal and sign a data use agreement.